CLINICAL TRIAL: NCT07367750
Title: Implementation of a Self-Management Support Program Among People With Kidney Transplant and Cancer Survivors in Israel: Testing Feasibility and Effects
Brief Title: Testing the Feasibility of a Self-Management Support Program for Patient With Chronic Diseases in Israel
Acronym: CDSMP-IL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Galit Yogev-Seligmann, researcher, Senior Lecturer, University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0703-24-TLV; no funding (Other Grant/Funding Number: no funding)
Record Dates: First submitted 2025-09-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Disease; Kidney Transplantation; Cancer Survivorship
Keywords: Chronic Disease; Self-Management; CDSMP; Kidney; Transplantation; Cancer Survivors
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDSMP Group (Experimental): Participants with chronic diseases (kidney transplant recipients or cancer survivors) will participate in the Chronic Disease Self-Management Program (CDSMP), a six-week online group intervention
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP)

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Program (CDSMP) — A structured, peer-led, six-week online intervention developed at Stanford University to enhance self-management skills in individuals with chronic conditions. Sessions include action planning, symptom management, medication adherence, healthy behaviors, and emotional coping.
  Other Names: Chronic Disease Self-Management Program(CDSMP)

SUMMARY:
This study explores an intervention to support people in Israel who are living with chronic health conditions such as cancer or after kidney transplantation. It focuses on a well-known international program called the Chronic Disease Self-Management Program (CDSMP), which was developed at Stanford University. The program helps individuals build confidence and skills to better manage their health, feel more in control, and improve their day-to-day quality of life.

Participants will take part in a six-week group program, delivered online, where they will learn practical strategies for managing symptoms like fatigue or pain, setting achievable health goals, communicating effectively with healthcare professionals, and staying active and engaged. The sessions are guided by trained facilitators and include support from others facing similar health challenges.

The study will involve surveys before and after the program, as well as a follow-up six months later, to understand how the program may have helped participants. Some participants will also be invited to share their experiences in small discussion groups.

By testing this program in Israel, the researchers hope to learn how it can be adapted and offered more widely to help others living with chronic conditions.

DETAILED DESCRIPTION:
This mixed-methods pilot study aims to evaluate the feasibility, acceptability, and potential impact of implementing the Chronic Disease Self-Management Program (CDSMP) in Israel. The CDSMP is an internationally recognized, evidence-based intervention originally developed at Stanford University to support individuals living with chronic health conditions. It is designed to improve self-efficacy, promote health-enhancing behaviors, and reduce the personal and healthcare burden associated with chronic illness.

The study will be conducted among adults with chronic conditions, specifically kidney transplant recipients and cancer survivors, recruited from a major tertiary care center(tel aviv sourasky medical center). Participants will take part in a 6-week group-based intervention delivered online in weekly 2.5-hour sessions. The sessions are led by trained facilitators certified in the CDSMP protocol and emphasize collaborative learning and peer support.

The program covers a range of self-management topics, including symptom management (e.g., fatigue, pain, sleep disturbances), medication adherence, physical activity, healthy eating, emotional coping, and communication with healthcare professionals. Participants are encouraged to engage in weekly action planning, goal setting, and problem-solving.

Quantitative data will be collected using validated self-report instruments at three time points: before the intervention, immediately after, and six months post-completion. These assessments will examine patient activation, engagement in health behaviors, symptom burden, and health-related quality of life.

In parallel, qualitative data will be gathered through focus groups with a subset of participants to capture their experiences and perspectives on the program. These discussions will explore perceived benefits, barriers to participation, and the program's impact on day-to-day functioning. Thematic analysis will be performed to identify key insights that may inform future adaptations and implementation strategies.

Findings from this pilot study will inform the potential for broader integration of the CDSMP into Israel's healthcare system and identify any cultural or operational adjustments needed for local relevance and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Diagnosed with at least one chronic disease (as documented in the medical record)
* Community-dwelling
* Fluent in Hebrew

Exclusion Criteria:

* Documented cognitive impairment
* Diagnosis of major depression or other psychiatric disorder (based on self-report or medical records)
* Hospitalization in the past 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM-13) | Baseline, immediately post-intervention, 6-month follow-up
  The Patient Activation Measure (PAM-13) is a validated self-report questionnaire that assesses individuals' knowledge, skills, and confidence in managing their health. Higher scores reflect greater activation and self-management ability.
health-related behaviors | Baseline, immediately post-intervention, 6-month follow-up
  Assessed using a custom self-report questionnaire developed by the research team, covering physical activity, nutrition, medication adherence, and use of health services.
chronic disease symptom burden | Baseline, immediately post-intervention, 6-month follow-up
  Evaluated using the Self-Management Resource Center (SMRC) symptom survey, which includes ratings of fatigue, pain, emotional distress, sleep, depression, anxiety, and social isolation.
health-related quality of life (EQ-5D) | Measured by the EQ-5D instrument, which assesses five dimensions of functioning and includes a global self-rated health visual analogue scale.
  Baseline, immediately post-intervention, 6-month follow-up

SECONDARY OUTCOMES:
Themes from focus group analysis regarding participant experience | through study completion, an average of 6-month
  Semi-structured focus groups will be conducted with a subset of participants to explore their perceptions of the program's relevance, usefulness, cultural fit, and overall impact on daily life. Audio recordings will be transcribed and analyzed thematically using a structured multi-stage coding process.
Perceived facilitators and barriers to self-management | through study completion, an average of 6-month
  Identified from qualitative data in focus group discussions. Participants will describe what helped or hindered their ability to engage in self-management behaviors following the intervention.
Participant suggestions for improving the CDSMP | through study completion, an average of 1 year
  Within one month after program completion

CONTACTS AND LOCATIONS:
Overall Officials: Galit Yogev-Seligmann, Principal Investigator — University of Haifa
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy considerations and the sensitive nature of the self-reported health and behavioral data collected. No plans for data sharing have been established at this time.